CLINICAL TRIAL: NCT01071967
Title: Effect of a Longitudinal, Multifactorial Community-based Nursing Intervention on Mortality in Chronically Ill Older Adults
Brief Title: Effect of a Community-based Nursing Intervention on Mortality in Chronically Ill Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Health Quality Partners (Other)
Collaborators: Centers for Medicare and Medicaid Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 95-C-91360/3-01
Record Dates: First submitted 2009-12-16; First posted 2010-02-19 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Heart Failure; Coronary Disease; Diabetes Mellitus; Asthma; Hypertension; Hypercholesterolemia
Keywords: Community Health Nursing; Nursing Care Management; Aged; Aged, 80 and over; Health Services for the Aged; Geriatric Nursing; Geriatric Assessment; Longevity; Mortality
MeSH Terms: conditions — Heart Failure; Coronary Disease; Diabetes Mellitus; Asthma; Hypertension; Hypercholesterolemia | interventions — Disease Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Community-based nurse care management (Experimental): Participants randomized to receive the intervention worked with a nurse care manager who provided them with a comprehensive set of geriatric and chronic disease preventive services.
  Interventions: Other: Community-based nurse care management
- Usual care (No Intervention): Participants randomized to the control group received usual care without the involvement of a nurse care manager.

INTERVENTIONS:
Other: Community-based nurse care management — The community-based nurse care management program developed by Health Quality Partners uses nurses working in the community to provide the following integrated set of services to older adults with chronic illness over the long term in order to prevent avoidable complications of their diseases and aging; geriatric assessment, care coordination, health education, self-management coaching, weight management, physical activity, gait and balance training, medication adherence, care transition support, ongoing monitoring and symptom detection, collaborative problem solving with patients, families and health care providers.
  Other Names: Health Quality Partners; Medicare Coordinated Care Demonstration; Care Coordination; Disease Management
  Arms: Community-based nurse care management

SUMMARY:
Care coordination, disease management, geriatric care management, and preventive programs for chronically ill older adults vary in design and their impact on long-term health outcomes is not well established. This study investigates whether a community-based nursing intervention improves longevity and impact on cardiovascular risk factors in this population. The results reflect the impact of one of the study sites (Health Quality Partners) selected by the Centers for Medicare and Medicaid Services (CMS) to participate in the Medicare Coordinated Care Demonstration, a national demonstration designed to identify promising models of care coordination for chronically ill older adults. The study began in April 2002.

DETAILED DESCRIPTION:
The community-based nursing care management model developed by Health Quality Partners represents a comprehensive set of integrated preventive and monitoring services designed for older adults living with chronic diseases. The individual programs and services integrated within the model were selected on the basis of previously demonstrated evidence of effectiveness. The model is delivered in the communities in which participants reside. Care is delivered through in person contacts, (1 to 1 and group) as well as by telephone. In person contacts occur in the home, in readily accessible community and faith-based organizations, health facilities, or the offices of Health Quality Partners. Efforts are made to contact participants in the intervention group at least monthly with care continued until death, voluntary disenrollment, mandatory disenrollment due to changes in insurance coverage, relocation out of the service area, or change in long term level of care (e.g., nursing home placement, hospice).

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years and older
* Medicare Part A and B traditional, fee for service insurance coverage
* One or more of the following chronic conditions:
* Heart failure
* Coronary Disease
* Diabetes mellitus
* Asthma
* Hypertension
* Hypercholesterolemia
* A Geriatric Risk Stratification Level of 2 or more based on a pre-enrollment screening tool
* Geriatric Risk Stratification Level changed in Sep 2006 to a Level of 3 or more
* Willingness of the participant's primary care provider to collaborate

Exclusion Criteria:

* Amyotrophic lateral sclerosis
* Alzheimer's disease
* Dementia
* Diagnosis or history of cancer (other than skin) in the past 5 years
* End-stage renal disease
* Life expectancy on enrollment less than 6 months
* HIV or AIDS
* Huntington's disease
* Organ transplant candidate
* Psychosis or schizophrenia
* Resident of or imminent plan for long-term nursing home placement
* Seasonal relocation outside of the area for more than 4 weeks per year
* Anyone receiving service from Health Quality Partners in the past

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2002-04; Primary Completion 2014-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | within 5 years of enrollment

SECONDARY OUTCOMES:
Blood pressure control | within 5 years of enrollment
Total cholesterol control | within 5 years of enrollment
Low density cholesterol control | within 5 years of enrollment
Triglycerides control | within 5 years of enrollment
Weight control | within 5 years of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth D Coburn, MD, MPH, Principal Investigator — Health Quality Partners
Locations (1):
- Health Quality Partners, Doylestown, Pennsylvania, United States

REFERENCES:
- [Background] Peikes D, Chen A, Schore J, Brown R. Effects of care coordination on hospitalization, quality of care, and health care expenditures among Medicare beneficiaries: 15 randomized trials. JAMA. 2009 Feb 11;301(6):603-18. doi: 10.1001/jama.2009.126. PMID 19211468
- [Background] Brown R, Peikes D, Chen A, Schore J. 15-site randomized trial of coordinated care in Medicare FFS. Health Care Financ Rev. 2008 Fall;30(1):5-25. PMID 19040171
- [Background] Bott DM, Kapp MC, Johnson LB, Magno LM. Disease management for chronically ill beneficiaries in traditional Medicare. Health Aff (Millwood). 2009 Jan-Feb;28(1):86-98. doi: 10.1377/hlthaff.28.1.86. PMID 19124858
- [Derived] Coburn KD, Marcantonio S, Lazansky R, Keller M, Davis N. Effect of a community-based nursing intervention on mortality in chronically ill older adults: a randomized controlled trial. PLoS Med. 2012;9(7):e1001265. doi: 10.1371/journal.pmed.1001265. Epub 2012 Jul 17. PMID 22815653
- See also: Health Quality Partners — http://www.hqp.org
- See also: Related ClinicalTrials.gov study — http://www.clinicaltrials.gov/ct2/show/NCT00627029?term=Medicare+Coordinated+Care+Demonstration&rank=1